CLINICAL TRIAL: NCT00000174
Title: Investigation Into Delay to Diagnosis of Alzheimer's Disease With Exelon (InDDEx)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: IA0012
Record Dates: First submitted 1999-10-29; First posted 1999-11-01 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-01

CONDITIONS: Alzheimer Disease; Cognition Disorders
Keywords: Mild cognitive impairment; Alzheimer's disease; Memory; Cholinergic agents; Cholinesterase inhibitors
MeSH Terms: conditions — Alzheimer Disease; Cognition Disorders; Cognitive Dysfunction | interventions — Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine

SUMMARY:
This phase IIIb trial is a prospective, randomized, double-blind, placebo-controlled, 36-month study comparing the length of time of progression from mild cognitive impairment (MCI) to a clinical diagnosis of Alzheimer's disease (AD) in subjects taking Exelon vs. placebo. Exelon is currently under review with the U.S. Food and Drug Administration as a treatment for Alzheimer's disease. The drug has been cleared for marketing in more than 40 countries for Alzheimer's disease to date, including all 15 member states of the European Union, New Zealand, Argentina, Brazil and Mexico.

Each subject with MCI will be randomly assigned to treatment with either Exelon or placebo. Subjects assigned to Exelon will receive 1.5 to 6.0 mg bid (twice daily) (3.0 to 12 mg/day) for the majority of the study. At every regular visit scheduled every three months, patients will be given basic efficacy and safety assessments. These assessments will include evaluation of adverse events, vital signs, activities of daily living, and clinical staging scales to determine if the subject may have converted to dementia.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 55-85 years, inclusive. Subjects older than 85 years may be eligible to participate, with approval of the designated study medical monitor.
* Are male or female without child-bearing potential (i.e., surgically sterilized [via bilateral tubal ligation,bilateral oophorectomy, or hysterectomy], at least one year postmenopausal, or using adequate birth control).
* Are cooperative, able to ingest oral medication, and willing to complete all aspects of the study.
* Will provide written informed consent prior to their participation in the study.
* Show evidence of mild cognitive impairment (MCI) by meeting all of the following criteria: Global CDR score = 0.5, NYU Delayed Paragraph Recall less than 9, 17-item HAM-D score less than 13, and HAM-D Item 1 (depressed mood) score =1.
* Have a friend or family member who is willing to participate in the study as an informant. The informant must see the subject at least once a week for several hours and be available to accompany the subject to the screening and baseline visits, and at a minimum, be accessible by telephone for other scheduled visits.

Exclusion Criteria:

* Advanced, severe, and unstable disease of any type that may interfere with primary and secondary variable evaluations including any medical condition that could be expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical or mental status of the subject to a significant degree or put the subject at special risk.
* Cognitive impairment sufficient to warrant a diagnosis of dementia.
* Met the DSM-IV and NINCDS-ADRDA criteria for AD.
* A clinical diagnosis of AD.
* A DSM-IV Axis 1 diagnosis. However, subjects with current depression are eligible after appropriate treatment of the depressive episode. A minimum of four weeks washout of antidepressant medication should occur prior to screening. Subjects with a prior history of depression (but not currently depressed) are allowed in the study.
* Fewer than four years of formal education.
* A documented history of transient ischemic attacks.
* Baseline MRI findings or CT-scan findings within a year of screening that are consistent with a process other than AD, e.g., stroke, tumor, brain trauma or hydrocephalus, that may contribute to the subject's MCI. Lacunae infarcts present in areas affecting cognition (entorhinal cortex, hippocampus, medial temporal lobe) will also exclude the subject from the study.
* A score of greater than 4 on the Modified Hachinski Ischemic Scale.
* A current diagnosis of any primary neurodegenerative disorder, e.g., Parkinson's disease.
* A current diagnosis of uncontrolled seizure disorder.
* A current diagnosis of active peptic ulceration.
* A current diagnosis of severe and unstable cardiovascular disease.
* A current diagnosis of sick-sinus syndrome or conduction deficits (sino-atrial block, second or third degree atrio-ventricular block).
* A current diagnosis of acute, severe, or unstable asthmatic conditions.
* A known exaggerated pharmacological sensitivity or hypersensitivity to drugs similar to Exelon or to other cholinergic compounds (e.g., pilocarpine, bethanechol, tacrine, velnacrine, donepezil, metrifonate, or physostigmine). Subjects who have experienced elevations in liver function test parameters on other cholinesterase inhibitors are still eligible.
* Taken any of the following substances: An investigational drug during the past four weeks; Metrifonate during the past three months; a drug or treatment known to cause major organ system toxicity during the past four weeks; other cholinergic drugs (e.g., donepezil, tacrine, succinylcholine-type muscle relaxants) during the past two weeks (topical pilocarpine will be permitted); antidepressant medication during the past four weeks.
* Participated in a previous clinical trial of Exelon.
* Clinically important laboratory abnormalities in serum B12, folate, or T3/T4 at screening. The subject should be excluded if peripheral neuropathy, macrocytic anemia, or myxedema is present.
* If screen values do not meet the absolutely exclusionary values given below but are still outside the normal reference range, treatment for folic acid/B12 deficiency or thyroid disorder, as appropriate, may be initiated or adjusted with re-evaluation of the subject within three months. Within these three months of treatment, the subject's cognitive condition must be clinically unchanged or worse for the subject to be acceptable. Once accepted, the subject must remain on the appropriate treatment throughout the study.
* Exclude if T3 uptake is less than 19%; T4 less than 2.9 ((g/dL); free T4 index is less than 0.8
* Exclude if folate less than 1.7 ng/ml (normal range greater than 1.9)
* Exclude if B12 less than 100 pg/ml (normal range greater than 200)
* A positive rapid plasmin reagin test followed up by a positive serological test for syphilis.
* A disability that may prevent the subject from completing all study requirements (e.g., blindness, deafness, severe language difficulty).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ferris, PhD, Principal Investigator — NYU Langone Health
Locations (15):
- United States (15):
  - Medici Research Centers, Peoria, Arizona
  - University of California, Irvine, Orange, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Neuromedical Research Institute (Offices in Ft. Lauderdale, Miami Beach and Boca Raton), Fort Lauderdale, Florida
  - Miami Research Associates, Miami, Florida
  - Center for Clinical Trials and Research, Venice, Florida
  - Indiana University Alzheimer's Center, Indianapolis, Indiana
  - St. Louis University, St Louis, Missouri
  - Alzheimer's Research Corporation, Lakewood, New Jersey
  - NYU Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Pahl Brain Associates, P.C., Oklahoma City, Oklahoma
  - Clinical Studies, Ltd., Philadelphia, Philadelphia, Pennsylvania
  - St. Paul Medical Center, Dallas, Texas
  - University of Washington, Seattle, Seattle, Washington

REFERENCES:
- [Derived] Feldman HH, Ferris S, Winblad B, Sfikas N, Mancione L, He Y, Tekin S, Burns A, Cummings J, del Ser T, Inzitari D, Orgogozo JM, Sauer H, Scheltens P, Scarpini E, Herrmann N, Farlow M, Potkin S, Charles HC, Fox NC, Lane R. Effect of rivastigmine on delay to diagnosis of Alzheimer's disease from mild cognitive impairment: the InDDEx study. Lancet Neurol. 2007 Jun;6(6):501-12. doi: 10.1016/S1474-4422(07)70109-6. PMID 17509485
- See also: The Alzheimer's Disease Education and Referral (ADEAR) Center is a service of the National Institute on Aging (NIA). — http://www.alzheimers.org